CLINICAL TRIAL: NCT03970941
Title: Two-stage Treatment of Large Bone Defects With Cerament® G and Cerament® V Plus Auto and/or Allograft Using the Masquelet Technique as Salvage Therapy After Bone Resection in Patients With Septic Pseudarthrosis
Acronym: EVIDENCE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0084
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Pseudarthrosis
MeSH Terms: conditions — Pseudarthrosis | interventions — Cost-Benefit Analysis; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CERAMENT: Patients having a septic pseudarthrosis managed with two-stage treatment (Masquelet Technique) with CERAMENT®.
  Interventions: Other: Cost evaluation; Other: Questionnaire
- NO CERAMENT COMPARATIVE COHORT: Patients having had a septic pseudarthrosis managed with two-stage treatment (only Masquelet Technique) without CERAMENT®.
  Interventions: Other: Cost evaluation

INTERVENTIONS:
Other: Cost evaluation — The cost for the hospital of the strategy of management will be evaluated.
Other: Questionnaire — The quality of life of patients will be measured.
  Groups: CERAMENT

SUMMARY:
Septic pseudarthrosis of long bones are complications that can unfortunately occur after the consolidation of a fracture and some situations present risks of superinfection, persistent infection or mechanical failure (30-40% risk of complications) that can lead to amputation.

A possible saving situation used by CRIOAC ("Centre de Référence des Infections Ostéo-Articulaires Complexes") is the use of a bone substitute impregnated with an antibiotic allowing a high local concentration of this antibiotic.

The aim of this study is to evaluate the cost of management of septic pseudarthrosis with two-stage treatment and CERAMENT® and the quality of life for this patients.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old
* Diagnosis of septic pseudarthrosis
* septic pseudarthrosis managed by the surgical technique using the CERAMENT bone substitute combined with an autograft / allograft by the Masquelet technique OR, for the comparative cohort: septic pseudarthrosis on long bone previously managed by the masquelet method without CERAMENT®
* Medico-surgical management within the CRIOAC ("Centre de Référence des Infections Ostéo-Articulaires Complexes") of the Croix-Rousse hospital in Lyon
* Patient who was informed and did not object to participate in the study

Exclusion Criteria:

* Patient with a disability (deafness, language disorders) or whose mental or cognitive state does not allow to be informed and to express his opposition if necessary.
* Patient with a disability (deafness, language impairment) or whose mental or cognitive state does not allow to understand the questions in the quality of life questionnaire
* Patient participating in another quality of life study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients having / having had a septic pseudarthrosis manage with two stage exchange (Masquelet technique)
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Cost evaluation | 24 months maximum
  Estimation of the cost of care from the point of view of the hospital This estimation will be measured at the end of patient follow-up (usually between 12 and 24 months after antibiotic therapy disruption)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Référence des Infections Ostéo-Articulaires complexes (CRIOAc) - Hôpital de la Croix-Rousse, Lyon, France

IPD SHARING:
Plan to Share IPD: No